CLINICAL TRIAL: NCT04632810
Title: The Norwegian LIPODIET Study: Effect of Ketosis on Pain and Quality of Life in Patients With Lipedema
Brief Title: Effect of Ketosis on Pain and Quality of Life in Patients With Lipedema
Acronym: Lipodiet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93888
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lipedema
Keywords: Diet therapy; Ketosis; Pain; Weight loss
MeSH Terms: conditions — Lipedema; Ketosis; Pain; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic low energy diet (Experimental): Ketogenic low energy diet for 8 weeks
  Interventions: Other: Ketogenic low energy diet
- non-Ketogenic low energy diet (Active Comparator): non-Ketogenic low energy diet for 8 weeks
  Interventions: Other: non-ketogenic low energy diet

INTERVENTIONS:
Other: Ketogenic low energy diet — Participants will follow a low energy diet, with 1200 kcal per day. Carbohydrates 75g (25E%), protein 60 g (20E%), fat 73 g (55E%) in 8 weeks
  Arms: Ketogenic low energy diet
Other: non-ketogenic low energy diet — Participants will follow a low energy diet, with 1200 kcal per day. Carbohydrates 180g (60E%), protein 60 g (20E%), fat 27 g (20E%), in 8 weeks
  Arms: non-Ketogenic low energy diet

SUMMARY:
Lipedema is a female progressive fat disorder, characterized by a symmetrical increase in subcutaneous adipose tissue in the lower extremities with the exception of the waist. The condition is often misdiagnosed and underdiagnosed. The etiology is poorly understood. Affects about 11% of all women and may lead to pain and immobility. The pathophysiology may be related to sex hormones and inflammatory response. Lipedema fat has been reported not to respond to lifestyle changes or bariatric surgery, both in terms of weight loss and symptom reduction; including pain and quality of life. Clinical research on the effect of dietary interventions on lipedema does not exist, but a pilot study with a ketogenic diet showed a significant reduction in pain regardless of weight loss. The aim of the research project will be to investigate whether a ketogenic diet can be a treatment option for patients with lipedema. Therefore, a randomized controlled trial will be conducted to compare the effects of two diets. 1) energy-restricted ketogenic diet and 3) energy-restricted low-fat non-ketogenic diet for 8 weeks. Pain and quality of life will be mesured at start and immediately after the intervention. The hypothesis is that a ketogenic diet may reduce pain and improve quality of life.

DETAILED DESCRIPTION:
Study design RCT comparing a low-energy ketogenic diet to a non-ketogenic low-energy diet (non-keto) in females with lipedema. This study was approved by the Reginal Ethical Committee (REK 93888) All participants have to provided written informed consent in line with the Helsinki Declaration, before entering the study. Participants will be randomized by block randomization with stratification by BMI categories.

Study population Females diagnosed with lipedema, aged 18-75 years old, and a BMI between 30-45 kg/m2, will be invited to participate in this study. Participants had to be diagnosed with lipedema by physiotherapists before inclusion. Inclusion criteria includs weight stability for the last three months (±3 kg).

Dietary interventions Diets were matched for energy (1200 kcal/day) and protein, but differed in carbohydrate (CHO) and fat content.

The dietary plans are adjusted with respect to food preferences, intolerances, and allergies. The participants will be asked not to change their physical activity levels throughout the study period.

Compliance Participants will have weekly follow-ups. Participants will be asked to fill out daily food records throughout the intervention period.

Ketostix will be used in the weekly follow-ups to measure urinary acetoacetate (AcAc). If the participants in the keto group were outside of ketosis, or participants in the non-keto group in ketosis, >2 times throughout the study period, they were excluded from the per-protocol (PP) analysis.

Outcome variables

The following variables were assessed at baseline and at the end of the intervention:

Anthropometrics and body composition Height and weight will be measured at baseline. Body composition will be assessed in fasting state with Bioelectrical Impedance Analysis before and after the intervention..

Pain Pain will be assessed with the brief Pain Inventory. The participants rated their pain in a numerical rating scale (NRS), where 0 = no pain and 10 = Worst imaginable pain. The BPI assesses pain intensity: strongest pain, weakest pain, average pain, pain now, pain severity score using an average of pain intensity domains, and pain inference from daily activities, mood, walking, regular work, relationships, sleep and life joy. A pain inference score is also computed as the average of all pain inference domains.

Three different questionnaires are used to assess Quality of life. RAND-36. The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) q and the Lymphoedema Quality of Life (LYMQOL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lipedema by skilled physical therapists
* Body mass index > 30kg/m2 and < 45kg/m2
* Stable weight over the last three months (+2-3kg)
* Not currently dieting to lose weight
* Willing to meet for follow-ups every second week during the intervention
* Willing to sign an informed consent before entering the study

Exclusion Criteria:

* Pregnant or breast feeding
* History of infectious diseases
* Medication known to affect obesity
* Enrolled in any other obesity treatment
* Having had bariatric surgery.
* Kidney disease is excluded
* History of psychological disorders
* Not mastering a Scandinavian language
* Being mentally disabled
* Malign disease
* Diabetes
* Any disease that leads to dietary advice that is not consistent with intervention advice

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | 8 weeks
  A difference in mean pain score of 2 units on a continuous scale from 0 to 10 on a visual analog scale (VAS) is considered clinically interesting
change in quality of life | 8 weeks
  Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Siren Nymo, PhD, Principal Investigator — Nord-Trøndelag Hospital Trust, Namsos Hospital, Clinic of Surgery; Hallvard Græslie, md, Study Director — Nord-Trøndelag Hospital Trust, Namsos Hospital, Clinic of Surgery
Locations (2):
- Norway (2):
  - Levanger Hospital, Nord-Trøndelag Hospital Trust, Levanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundanes J, Nes VF, Aakervik O, Ryan L, Hansson P, Rokstad AM, Martins C, Nymo S. Changes in Cytokines and Fibrotic Growth Factors after Low-Carbohydrate or Low-Fat Low-Energy Diets in Females with Lipedema. Curr Dev Nutr. 2025 Feb 20;9(3):104571. doi: 10.1016/j.cdnut.2025.104571. eCollection 2025 Mar. PMID 40125475
- [Derived] Lundanes J, Garseth M, Taylor S, Crescenzi R, Pridmore M, Wagnild R, Hyldmo AA, Martins C, Nymo S. The effect of a low-carbohydrate diet on subcutaneous adipose tissue in females with lipedema. Front Nutr. 2024 Nov 7;11:1484612. doi: 10.3389/fnut.2024.1484612. eCollection 2024. PMID 39574523
- [Derived] Lundanes J, Storlilokken GE, Solem MS, Dankel SN, Tangvik RJ, Odegard R, Holst JJ, Rehfeld JF, Martins C, Nymo S. Gastrointestinal hormones and subjective ratings of appetite after low-carbohydrate vs low-fat low-energy diets in females with lipedema - A randomized controlled trial. Clin Nutr ESPEN. 2025 Feb;65:16-24. doi: 10.1016/j.clnesp.2024.11.018. Epub 2024 Nov 19. PMID 39566600